CLINICAL TRIAL: NCT03119870
Title: Structure-function Relationships Within the Cingulate Cortex
Brief Title: Organization of the Cingulate Cortex
Acronym: EEG-Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0659
Record Dates: First submitted 2017-03-09; First posted 2017-04-19 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: fMRI; EEG; behavior; cingulate cortex
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Each subject will conduct 3 sessions, i.e. a training session, an anatomical MRI session and an EEG session. The first session will be to train the subject to carry out the different behavioral tasks that he will then have to perform during the session of EEG.
  Interventions: Other: Train; Other: MRI; Other: EEG

INTERVENTIONS:
Other: Train — Each subject will be trained to perform a trial-error learning task. In this task, three visual stimuli will be presented to the subject. The subject will have to find by trial-error, the one associated with positive feedback, the other stimuli being associated with negative feedback (search period). Once the stimulus is associated with positive feedback, the subject will perform a period of repetition during which he will choose the stimulus associated with positive feedback. Two variants of the task will be used: a variant in which feedback will be visual (ie positive feedback = green square, negative feedback = red square) and a variant in which feedback will be fruit juice (ie positive feedback = Fruit juice (but less than 2ml), negative feedback = no volume or small volume of fruit juice).
Other: MRI — Once the tasks are learned, each subject will participate in an MRI session during which an anatomical scan will be obtained. For each task, the time of presentation of the stimuli will be 2s. During this time, the subject should indicate his choice of stimulus. After a delay of 2s, feedback will be presented for 1s. Each test shall be separated by an inter-test delay of 3s. The presentation of the stimuli and the control of the answers will be managed by the E-prime or Presentation software.
Other: EEG — Once the tasks are learned, each subject will participate in an MRI session during which an anatomical scan will be obtained and then an EEG session during which he will perform the task learned.For each task, the time of presentation of the stimuli will be 2s. During this time, the subject should indicate his choice of stimulus. After a delay of 2s, feedback will be presented for 1s. Each test shall be separated by an inter-test delay of 3s. The presentation of the stimuli and the control of the answers will be managed by the E-prime or Presentation software.

SUMMARY:
Efficient evaluation and monitoring of actions and outcomes are a key feature of primates' efficient adaptive cognition. Deficits in evaluating one's own actions and their consequences is a key feature of prominent disorders such as obsessive compulsive disorders (OCD), schizophrenia, and anxiety. The Investigators know that these evaluative processes implicate medial structures of the brain that are related both to old limbic functions and to more recently evolved higher executive functions. Brain potentials related to performance monitoring have attracted a lot of interest in cognitive neuroscience but also in the clinical domain because they appear to be altered in different neurological or psychiatric disorders, such as schizophrenia, OCD, or anxiety, and could become biomarkers of pathologies. But the neural sources of these markers are not fully determined and are currently highly debated. In addition, our work suggests that non pathological factors, such as normal morphological cortical variations, could affect those markers. Understanding performance monitoring, acting directly on medial cortex, or using electrophysiological markers in clinic are thus currently problematic and challenging. This is mostly because structure-function relationships in the medial wall are ill defined for historical, conceptual, and methodological reasons. Importantly, although individual variability of brain morphology impedes precise assessment of structure function relationships, this variability is almost never taken into account. EEG-Feedback aims to resolve these issues by evaluating the consequences of individual variability in cingulate cortex morphology on 1) surface EEG markers of feedback monitoring and 2) functional connectivity patterns thanks to resting-state fMRI.

ELIGIBILITY:
Inclusion Criteria:

* being able to provide a writen consent form
* having a social insurance
* have a normal vision (with or without corrections)
* Right-handed

Exclusion Criteria:

* Subjects with MRI contraindications (e.g. pacemaker, claustrophobia, metal in the body, etc…).
* Subjects must be willing to be advise in case of discovery of brain abnormality.
* No history of known neurological or psychiatric illness
* Pregnant or nursing women
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights or liberty, as well as legal persons protected by law

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2013-09-06 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Resting state fMRI data | 3 years
  BOLD signal will be analyzed in the low frequency band (0.1-0.01Hz). Images must be not too much distorted to allow data analysis. As such, if a subject moved too much (translation>10mm; rotation>5°) the corresponding data will be excluded from the analysis.
EEG data | 3 years
  If recordings are too noisy (if only <30% of trials survive the denoising process), subject will be excluded from final analysis.
Behavioral data in the EEG experiment | 3 years
  Performance in the task will be assessed. If performance in the task is <80%, subjects will be excluded in the final analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Christian SCHEIBER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Groupement Hospitalier Est, Bron, France